CLINICAL TRIAL: NCT01710280
Title: Palmitic Acid in the Sn-2 Position of Triacylglycerols and Postprandial Lipemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Wendy Hall, Lecturer in Nutritional Sciences, King's College London
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRIS
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Healthy Men; Raised Fasting Plasma Triacylglycerol Concentrations
Keywords: Lipemia; Vascular function; Blood pressure
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Native palm olein (Active Comparator): 75 g native palm olein
  Interventions: Dietary Supplement: High-fat meal containing native palm olein
- Interesterified palm olein (Experimental): 75 g interesterified palm olein
  Interventions: Dietary Supplement: High-fat meal containing interesterified palm olein

INTERVENTIONS:
Dietary Supplement: High-fat meal containing native palm olein
  Arms: Native palm olein
Dietary Supplement: High-fat meal containing interesterified palm olein
  Arms: Interesterified palm olein

SUMMARY:
The purpose of this study is to determine whether high-fat meals rich in palmitic acid in the sn-2 position decrease lipaemia in men aged 40-70 y with higher than optimal fasting triacylglycerol concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Non-smokers
* Aged 40-70 years
* Fasting TAG concentrations ≥1.5 mmol/L.

Exclusion Criteria:

* Reported history of CVD (myocardial infarction, angina, venous thrombosis, stroke), impaired fasting glucose/uncontrolled type 2 diabetes (or fasting glucose ≥ 6.1 mmol/L), cancer, kidney, liver or bowel disease.
* Presence of gastrointestinal disorder or use of drug, which is likely to alter gastrointestinal motility or nutrient absorption.
* History of substance abuse or alcoholism (previous weekly alcohol intake >60 units/men)
* Current self-reported weekly alcohol intake exceeding 28 units
* Allergy or intolerance to any component of test meals
* Unwilling to restrict consumption of any source of fish oil for the length of the study
* Weight change of >3kg in preceding 2 months
* Body Mass Index <20 and >35 kg/m2
* Fasting blood cholesterol > 7.8 mmol/L
* Current cigarette smoker.
* Current use of lipid lowering medication

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Incremental AUC (change from baseline in overall response) for plasma triacylglycerol concentrations | 1-6 h post-meal

SECONDARY OUTCOMES:
Incremental AUC for plasma non-esterified fatty acid concentrations | 1-6 h post-meal
Changes from baseline in digital volume pulse | 2,4,5,6 h post-meal
Changes from baseline in blood pressure | 2,4,5,6 h post-meal

OTHER OUTCOMES:
Incremental AUC for plasma total cholesterol concentrations | 1-6 h post-meal

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes & Nutritional Sciences Division, King's College London., London, United Kingdom

REFERENCES:
- [Background] Sanders TA, Filippou A, Berry SE, Baumgartner S, Mensink RP. Palmitic acid in the sn-2 position of triacylglycerols acutely influences postprandial lipid metabolism. Am J Clin Nutr. 2011 Dec;94(6):1433-41. doi: 10.3945/ajcn.111.017459. Epub 2011 Oct 26. PMID 22030225
- See also: Primary publication — http://www.ncbi.nlm.nih.gov/pubmed/25103522